CLINICAL TRIAL: NCT02488499
Title: Addressing Behaviour and Treatment Effectiveness Project (A.B.A.T.E. Project)
Acronym: ABATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Ontario Mental Health Foundation (Other Government)
Responsible Party: Principal Investigator, Brendan Andrade, Clinician-Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 091/2010-03
Record Dates: First submitted 2015-06-24; First posted 2015-07-02 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Disruptive Behavior Disorder
Keywords: Disruptive Behaviour Disorder; Psychosocial; Group Treatment
MeSH Terms: conditions — Attention Deficit and Disruptive Behavior Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Individualized Treatment (Active Comparator): Individualized Treatment: 15 sessions of individualized treatment (i.e., parent-child) that target areas of presenting concern identified during assessment. These may include social problem-solving, emotion regulation, parent-child difficulties.
  Interventions: Behavioral: Individualized Treatment
- Coping Power (Experimental): Coping Power: 15 sessions of concurrent parent and child group treatment. The child group focuses on developing problem-solving and emotion regulation skills. The parent group focuses on developing parenting skills and problem-solving strategies to manage and reduce their children's disruptive behaviour.
  Interventions: Behavioral: Coping Power

INTERVENTIONS:
Behavioral: Coping Power — 15 sessions of concurrent parent and child group treatment
  Arms: Coping Power
Behavioral: Individualized Treatment — 15 sessions of individualized child and parent treatment
  Arms: Individualized Treatment

SUMMARY:
This study investigates the effectiveness of a clinic-adapted version of the Coping Power program compared to individualized child and family treatment for children with disruptive behaviour and their parents.

DETAILED DESCRIPTION:
This project compares the short- and long-term effectiveness of a clinic-adapted manualized group treatment (i.e., Coping Power; CP) to individualized child and family treatment for children aged 9 - 12 with disruptive behaviour. Children and their parents who meet criteria and agree to participate in the project are randomly assigned to either the CP condition or the Individualized treatment condition. In the CP condition, children and caregivers are asked to participate in two separate but complimentary 15-session groups. Child groups target development of children's emotional and cognitive problem solving skills and caregiver groups facilitate cognitive and behavioural parenting skills. In the Individualized treatment condition children and caregivers are asked to participate in 15 one-hour individual and family treatment sessions tailored by the clinician to address the children and parent's presenting concerns. Measurement of behaviour and emotional functioning is done pre- post- and at 6-months following treatment.

ELIGIBILITY:
Inclusion Criteria:

* Parents provide free and informed consent and children assent to participate in the research, complete measures, and participate in either Coping Power or individualized treatment.
* Parents report symptoms consistent with clinical diagnoses of Oppositional Defiant Disorder or Conduct Disorder on the Diagnostic Interview Schedule for Children - DSM IV or parents and/or teacher report at or above a T-score of 60 (93rd percentile; borderline clinically severe range) on the Externalizing Behavior composite scale on the Behavior Assessment for Children - 2nd edition.
* Parents or teachers report clinically severe impairment in social, family, peer or overall functioning demonstrated by scores in the clinical range on the parent or teacher completed Impairment Rating Scale.
* The child's cognitive functioning is at or above a standard score of 80 (Borderline Range) on the verbal and/or nonverbal scales on the Kaufman Brief Intelligence Task - 2.

Exclusion Criteria:

* Evidence of Autism Spectrum Disorder or Asperger's Disorder as reported by parent, teacher or physician referral (if available).

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 172 (Actual)
Dates: Start 2010-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Conduct Problems scale score measured by the Strengths and Difficulties Questionnaire | Change from Baseline Conduct Problems at 15-weeks and at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Brendan F Andrade, Ph.D., Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- [Background] Lochman JE, Powell N, Boxmeyer C, Andrade B, Stromeyer SL, Jimenez-Camargo LA. Adaptations to the coping power program's structure, delivery settings, and clinician training. Psychotherapy (Chic). 2012 Jun;49(2):135-42. doi: 10.1037/a0027165. PMID 22642521
- [Background] Wells, K. C., Lochman, J. E., & Lenhart, L. A. (2008). Coping Power Parent Group Program: Facilitator Guide. New York: Oxford University Press.
- [Background] Wells, K. C., Lochman, J. E., & Lenhart, L. A. (2008b). Coping Power: Facilitators Guide. New York: Oxford Press
- [Background] Lochman JE, Wells KC. The coping power program for preadolescent aggressive boys and their parents: outcome effects at the 1-year follow-up. J Consult Clin Psychol. 2004 Aug;72(4):571-8. doi: 10.1037/0022-006X.72.4.571. PMID 15301641
- See also: CAMH Research — http://www.camh.net/research